CLINICAL TRIAL: NCT02750956
Title: Effect of Non-surgical Periodontal Treatment on Gingival Crevicular Fluid and Serum Endocan, Vascular Endothelial Growth Factor-A and Tumor Necrosis Factor Alpha Levels
Brief Title: Endocan, VEGF and TNF-alpha Levels in Periodontal Disease and After Treatment
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, ÇİĞDEM COŞKUN TÜRER, Dr., Bulent Ecevit University
Other Study IDs: Endocan
Record Dates: First submitted 2016-04-19; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Periodontal Disease
Keywords: endocan protein; VEGF A; TNF-alpha; after treatment
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid and Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Periodontal healthy individuals
- Group 2: Patients with chronic periodontitis
  Interventions: Procedure: Non-surgical periodontal treatment
- Group 3: the same patients in group 2 after they had been treated with scaling and root planing (SRP) were considered as Group 3.
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Non-surgical periodontal therapy is an anti-infective therapy which includes both mechanical and chemotherapeutic approaches to minimize or eliminate microbial biofilm, the primary etiology of gingivitis and periodontitis
  Groups: Group 2; Group 3

SUMMARY:
The primer aim of the study was to determine serum and gingival crevicular fluid (GCF) endocan levels in periodontal diseases pathogenesis supported with vascular endothelial growth factor (VEGF) and tumor necrosis factor alpha (TNF-α) levels.

DETAILED DESCRIPTION:
The study consist of three groups: periodontally healthy individuals (group 1; n = 20), individuals with generalized chronic periodontitis (group 2; n = 20), the same patients with chronic periodontitis after they had been treated with scaling and root planing (SRP) were considered as Group 3. Clinical measurements were recorded; GCF and serum samples were obtained from each participant before and 6 weeks after therapy. Endocan, VEGF-A and TNF-α levels were measured by enzyme-linked immunosorbent assay.

ELIGIBILITY:
Group 1 Inclusion Criteria:

* No bone and attachment loss,
* GI=0, PPD≤3mm, CAL≤3mm
* Systematically healthy patients

Group 2 Inclusion Criteria:

* GI>1, PPD≥5mm, CAL≥5mm with alveolar bone loss radiographically.
* Systematically healthy patients

Exclusion Criteria:

* Aggressive Periodontitis,
* Oral pathologies,
* Patients with any other systemic diseases,
* Pregnant women and those in the lactation period,
* Patients with smoking habit and taking medication
* Patients received periodontal therapy in last 6 months

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Total of 40 individuals
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Endocan levels | 6 weeks
  Change after periodontal treatment

SECONDARY OUTCOMES:
VEGF levels | 6 weeks
  Change after periodontal treatment
TNF-alpha levels | 6 weeks
  Change after periodontal treatment

CONTACTS AND LOCATIONS:
Overall Officials: ÇİĞDEM COŞKUN TÜRER, Principal Investigator — BULENT ECEVIT UNIVERSITY FACULTY OF DENTISTRY DEPARTMENT OF PERIODONTOLOGY

IPD SHARING:
Plan to Share IPD: No